CLINICAL TRIAL: NCT05044585
Title: Evaluation of RDS MultiSense® in Desaturation Analysis and Effects of Hypoxia on Circulating Oxidative Stress and Mitochondrial Respiration in Healthy Volunteers
Brief Title: Evaluation of RDS MultiSense® in Desaturation Analysis in Healthy Volunteers
Acronym: HYPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Collaborators: Rhythm Diagnostic Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-001
Record Dates: First submitted 2021-08-26; First posted 2021-09-16 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Hypoxia
Keywords: vital signs; connected device; real-time monitoring; hypoxia; SpO2; non-invasive blood pressure; cardio-respiratory monitoring
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: prospective feasibility study,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Automated Monitoring System (Experimental): Two MultiSense® patches will be placed on each volunteer. The monitoring will last no more than 3 hours, during an induced and controlled hypoxia.
  Interventions: Other: Remote Automated Monitoring System

INTERVENTIONS:
Other: Remote Automated Monitoring System — The subject will be monitored with conventional monitoring devices as well as the MultiSense patch.

SUMMARY:
In this clinical study, the investigators will compare vital parameters measurements obtained using continuous data from reference monitors and continuous wireless MultiSense® monitoring patch in 30 healthy volunteers under induced and controlled hypoxia.

DETAILED DESCRIPTION:
The MultiSense® strip is a unique, band aid-sized, clinical signal quality, connected strip for real-time monitoring of cardio-respiratory parameters. The MultiSense® strip measures in real-time, remotely and continuously 11 clinical key-indicators by being attached to the patient thorax: ECG trace, heart rate, oxygen saturation, respiratory rate and relative respiration depth, pulse transit time, plethysmographic trace, perfusion index, skin temperature, physical activity and body position. Designed to be worn continuously for at least seven days, the patient can keep the patch during his sleep or in the shower.

The aim of this study is to determine the quality of measurements of arterial blood saturation (SpO2) provided by the MultiSense® system in comparison to measurements made with a reference Pulse Oximetry System under induced hypoxia, in terms of accuracy.

The study population includes 30 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 to 50 years of age.
* Subject able to receive and understand information related to the study and give written informed consent.
* Subject is a non-smoker or an ex-smoker (stopped smoking for at least 6 months).
* Subject demographics include a range of dark skin pigmentations, including at least 30% of the total pool, assessed by phototypes V and VI according to the Fitzpatrick scale (Questionnaire score between 28 and 40).
* Subject is healthy (assessed by a physical examination AND normal ECG AND absence of medical treatment except for the birth control pill).
* Subject authorizing the treatment of their personal data collected during the study (box checked in the consent form).
* Subject affiliated to the French social security system.

Exclusion Criteria:

* Subject with antecedent of allergies to adhesives or silicone or a skin disease that would preclude the use of an adhesive.
* Subject with an implantable device such as a pacemaker.
* Pregnant or lactating women (assessed by a negative ß-HCG test).
* Subject with a high-altitude stay during the previous 4 weeks (more than 1 week spent over 3,500 meters).
* Subject with Raynaud's syndrome.
* Subject in exclusion period (determined by a previous or a current study).
* Subject under guardianship or trusteeship.
* Subject under the protection of justice.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Determination of the quality of measurements of arterial blood saturation (SpO2) provided by the MultiSense® system in comparison to measurements made with a reference Pulse Oximetry System, in terms of accuracy. | from patch placement to patch removal, assessed up to 3 hours
  Accuracy is defined as an average measurement variation less than 3.5% of the mean value to the reference standard. The data for analysis will be equally distributed across the SpO2 range of 70-100%.

SECONDARY OUTCOMES:
Descriptive kinetic of circulating oxidative stress markers under hypoxia conditions | from patch placement to patch removal, assessed up to 3 hours
  comparison of circulating oxidative stress and plasma antioxidant activity markers in blood between hypoxia and normal oxygenation conditions by dosage of anion superoxide (µmol/min)
Descriptive kinetic of circulating oxidative stress markers under hypoxia conditions | from patch placement to patch removal, assessed up to 3 hours
  comparison of circulating oxidative stress and plasma antioxidant activity markers in blood between hypoxia and normal oxygenation conditions by dosage of lipids peroxidation (µg/mL)
Descriptive kinetic of circulating oxidative stress markers under hypoxia conditions | from patch placement to patch removal, assessed up to 3 hours
  comparison of circulating oxidative stress and plasma antioxidant activity markers in blood between hypoxia and normal oxygenation conditions by dosage of protein carbonylation (ng/mL)
Descriptive kinetic of circulating oxidative stress markers under hypoxia conditions | from patch placement to patch removal, assessed up to 3 hours
  comparison of circulating oxidative stress and plasma antioxidant activity markers in blood between hypoxia and normal oxygenation conditions by dosage of catalase (U/mg protein)
Descriptive kinetic of circulating oxidative stress markers under hypoxia conditions | from patch placement to patch removal, assessed up to 3 hours
  comparison of circulating oxidative stress and plasma antioxidant activity markers in blood between hypoxia and normal oxygenation conditions by dosage of superoxide dismutase (U/mg protein)
Descriptive kinetic of circulating oxidative stress markers under hypoxia conditions | from patch placement to patch removal, assessed up to 3 hours
  comparison of circulating oxidative stress and plasma antioxidant activity markers in blood between hypoxia and normal oxygenation conditions by dosage of glutathione (µmol/g protein)
Comparison of Mitochondrial respiration from PBMCs between hypoxia and normal oxygenation conditions. | from patch placement to patch removal, assessed up to 3 hours
  Mitochondrial respiration from PBMCs is assessed by high-resolution respirometry by analysis of the kinetic of the respirometry results and comparison between each hypoxia /post-hypoxia data point with the baseline.
To evaluate the impact of skin pigmentation on SpO2 determination by the MultiSense® solution. | from patch placement to patch removal, assessed up to 3 hours
  Comparison of the MultiSense® SpO2 performances with the reference between light and dark-pigmented subjects. Qualitative comparison of the raw PPG signal between light and dark-pigmented skin subjects.
To evaluate pulse transit time (PTT) as an indicator of blood pressure (BP) variation. | from patch placement to patch removal, assessed up to 3 hours
  Comparison of blood pressure variation measured by a standard cuff device with PTT variation measured by the MultiSense® acquisition system.
To evaluate the reliability of the respiration rate determined by the MultiSense® solution | from patch placement to patch removal, assessed up to 3 hours
  Determination of the quality of respiration rate provided by the MultiSense® patch in comparison to measurements made with reference medical devices in the hospital setting, in terms of accuracy. Accuracy is defined as an average measurement variation less than 5% of the respiration rate mean value to the reference standard.
To compare the quality of MultiSense® data from a patch worn on the chest and from a patch worn on the upper back in different body posture and to evaluate the impact of strip exact localization on the chest. | from patch placement to patch removal, assessed up to 3 hours
  Qualitative comparison of the raw PPG signal between the two patches location for each subject (chest and back). Comparison of the SpO2 derived by each MultiSense® patch to the reference during the resting period in different lying positions (supine, prone, left and right side).

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Geny, Pr, Principal Investigator — Physiology and Functional Exploration, NHC Strasbourg, France
Locations (1):
- Clinical Investigation Center & Physiology and Functional Explorations unit at NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No